CLINICAL TRIAL: NCT05252767
Title: Evaluation of an Intervention for Improving Patient Engagement in Perioperative Pain Management
Brief Title: Patient Engagement in Perioperative Pain Management Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00307176; R01CE003150 (NIH)
Record Dates: First submitted 2022-02-14; First posted 2022-02-23 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Pain, Postoperative; Opioid Use Disorder
Keywords: Patient engagement; Patient activation
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders; Patient Participation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A - Patient Engagement Tools (Experimental): Participants will be enrolled from the a pain management clinic. Participants randomized into the experimental cohort will receive access to a clinic brochure, clinic website, as well as 'My Pain Passport' and 'My Treatment Plan' tools.
  Interventions: Behavioral: Patient Engagement Tools
- Cohort B - Educational Guide (Sham Comparator): Participants randomized into the control cohort will receive a brief educational guide on general pain management.
  Interventions: Behavioral: Educational Guide

INTERVENTIONS:
Behavioral: Patient Engagement Tools — Experimental participants will receive the patient engagement tools or the educational guide after randomization. The participants in the experimental cohort will utilize the tools between visits with their clinic providers. During visits, clinic providers will review the completed tools with participants.
  Arms: Cohort A - Patient Engagement Tools
Behavioral: Educational Guide — Control participants will receive a brief educational guide about pain management.
  Arms: Cohort B - Educational Guide

SUMMARY:
Previously, the study team evaluated the implementation and effectiveness of the Johns Hopkins Perioperative Pain Program (PPP), which coordinates continuum of care for surgical patients on chronic opioid therapy throughout the perioperative period. Based on the findings of that project, the study team developed an educational intervention intended to improve patient engagement in perioperative pain management. In this project, the study team will formally implement a randomized controlled trial to evaluate the effectiveness of the intervention developed.

ELIGIBILITY:
Inclusion Criteria:

* All patients in Johns Hopkins Personalized Pain Program Clinic

Exclusion Criteria:

* Active suicidal ideation at study entry
* Primary psychotic disorder
* Non-English speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Patient engagement as assessed by a patient engagement survey | Time of each participant's standard of care clinic visit, up to 1 year from enrollment
  Patient engagement survey measures level of patient engagement on five-point Likert scale

SECONDARY OUTCOMES:
Opioid consumption as assessed by daily morphine milligram equivalents | Time of each participant's standard of care clinic visit, up to 1 year from enrollment
  Daily morphine milligram equivalents (MME) indicates potency of an opioid dosage compared to morphine
Pain level as assessed by the Brief Pain Inventory | Time of each participant's standard of care clinic visit, up to 1 year from enrollment
  Brief Pain Inventory assesses pain severity and impact of pain on functional status on 10-point scale (1=no pain, no interference and 10 = worst pain, complete interference)
Pain level as assessed by the Present Pain Intensity scale of the McGill Pain Questionnaire | Time of each participant's standard of care clinic visit, up to 1 year from enrollment
  Present Pain Intensity scale of the McGill Pain Questionnaire measures pain intensity on 4-point scale (0 = none, 3 = severe)
Pain level as assessed by the Pain Catastrophizing Scale | Time of each participant's standard of care clinic visit, up to 1 year from enrollment
  Pain Catastrophizing Scale measures level of pain catastrophizing (0 = not at all, 4 = all the time)
Functional status as assessed by the Insomnia Severity Index | Time of each participant's standard of care clinic visit, up to 1 year from enrollment
  Insomnia Severity Index measures severity of insomnia on five-point scale (0=none, 4=severe, were score of 0-7 indicates no clinically significant insomnia and score of 22-28 indicates clinical or severe insomnia)
Functional status as assessed by the 36-Item Short Form Health Survey | Time of each participant's standard of care clinic visit, up to 1 year from enrollment
  36-Item Short Form Health Survey measures overall health status (converted into 0-100 scale, were lower score indicates more disability)

CONTACTS AND LOCATIONS:
Overall Officials: Anping Xie, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No